CLINICAL TRIAL: NCT04561791
Title: Evaluation of Tethered Capsule Endomicroscopy as a Screening Tool for Barrett's Esophagus in the Primary Care Setting
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Guillermo J. Tearney, MD, PhD, FACC, FCAP, FNAI, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018P002403
Record Dates: First submitted 2020-08-11; First posted 2020-09-24 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Barrett Esophagus; Barrett's Esophagus Without Dysplasia; Barretts Esophagus With Dysplasia
Keywords: OCT; Optical Coherence Tomography; Endomicroscopy; Capsule Endomicroscopy; Tethered Capsule Endomicroscopy; TCE
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Feasibility of TCE & Prevalence of BE (Experimental): 1. Feasibility of using tethered capsule endomicroscopy as a screening method for Barrett's esophagus in the primary care practice environment
  2. Determine the prevalence of Barrett's esophagus in a primary care practice cohort at MGH
  Interventions: Device: Tethered Capsule Endomicroscopy

INTERVENTIONS:
Device: Tethered Capsule Endomicroscopy — Participants will be asked to swallow the TCE device. Participants may use mild numbing spray, and lubrication spray to help swallowing. Imaging will be conducted once the TCE device is past the pharynx. The TCE device will be advanced until the stomach and then slowly pull the TCE back up the esophagus. This may be repeated twice.

SUMMARY:
The investigators will conduct a large study in the primary care clinic to determine the feasibility of using tethered capsule endomicroscopy as a screening method for Barrett's esophagus (BE) in the primary care practice environment. The investigators are also determining the prevalence of Barrett's esophagus in a primary care practice cohort at MGH.

DETAILED DESCRIPTION:
The investigators have developed a tethered capsule OCT device intended as an inexpensive screening tool for BE. The capsule, which is attached to a thin, flexible tether, is reusable after being processed by a standard disinfection technique. Used without sedation, the capsule is swallowed by the participant and travels in the esophagus to the gastroesophageal junction (GEJ) via peristalsis. Cross-sectional microscopic OCT images of the entire esophagus are collected during transit. The total time needed for swallowing, imaging and retrieval does not exceed 10 minutes, with a total of 30 minutes for the procedure. The investigators have tested the feasibility and the tolerability of this new OCT screening technology in 250 procedures in healthy volunteers and participants with various esophageal diseases including BE. The procedure has been safe and well tolerated. High quality microscopic images of the esophagus have been obtained in 90% of the enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants registered as patients at the Assembly Row primary care practice, MGH Broadway Primary Care - Revere, or Pentucket Medical Associates
* 18 years or older
* Able to give informed consent
* Participants must have no food for 1 hour before the procedure

Exclusion Criteria:

* Participants older than 75 years.
* Participants with current symptoms of dysphagia
* Participants with gastro-intestinal strictures with a diameter less than 8mm, prior GI surgery (Esophageal and/or stomach surgeries), or history of intestinal Crohn's disease
* Pregnancy
* Participants scheduled for an urgent care visit for the following symptoms: fever, sore throat, upper respiratory infection symptoms, nausea, vomiting, diarrhea, abdominal pain, or other symptoms as per clinical staff discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Subject Tolerability of Tethered Capsule Endomicroscopy Swallow | During the single study visit (avg 30.mins), and before leaving, the participant will fill out the tolerability survey
  The study team will ask the participant about their comfort level throughout the procedure. Participants will be asked to score the tolerability of the procedure using a scoring system from 0-10. 0= the least tolerable, 10= the most tolerable. The title of the scale is Subject Tolerability Questionnaire.
Prevalence of Barrett's esophagus within the single Primary Care Practice cohort. | Imaging data is collected during the procedure, and analyzed within 1 year of collection.
  The PI will identify signs of Barrett's esophagus from the imaging data. This is a qualitative assessment performed by the PI, as this imaging technique is to novel to have standard quality grading.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D, PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No